CLINICAL TRIAL: NCT05810272
Title: The Impact of Postprandial 'Exercise Snacks' on Protein and Glucose Metabolism Following a Period of Step Reduction in Older Adults
Brief Title: Impact of Postprandial 'Exercise Snacks' on Protein and Glucose Metabolism Following a Period of Step Reduction in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Associate Professor in Muscle Physiology, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ESPEN
Record Dates: First submitted 2023-02-21; First posted 2023-04-12 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Inactivity, Physical; Aging; Healthy Aging; Sarcopenia; Muscular Atrophy; Neuromuscular Manifestations; Neurologic Manifestations; Nervous System Diseases; Atrophy; Pathological Conditions, Anatomical
Keywords: Skeletal Muscle; Step-Reduction; Aging; Anabolic Resistance; Physical Activity; Stable Isotopes
MeSH Terms: conditions — Sedentary Behavior; Sarcopenia; Muscular Atrophy; Neuromuscular Manifestations; Neurologic Manifestations; Nervous System Diseases; Atrophy; Pathological Conditions, Anatomical; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Habitual Activity (Other): Following three days of habitual activity, a metabolic trial will be completed wherein participants (10M/10F) will be assessed for their anabolic response to a protein-carbohydrate meal.
  Interventions: Behavioral: Metabolic Trial
- Step-Reduction (Experimental): Participants will undergo three days of reduced physical activity (<1,500 steps/day) prior to a metabolic trial to establish their anabolic response to a protein-carbohydrate meal.
  Interventions: Behavioral: Metabolic Trial; Behavioral: 15 sit-to-stands with calf raises

INTERVENTIONS:
Behavioral: Metabolic Trial — Participants will undergo a metabolic trial to assess for their anabolic response to a protein-carbohydrate meal.
Behavioral: 15 sit-to-stands with calf raises — Participants (n=10; 5F/5M) will be randomized to perform 15 sit-to-stands with calf raises every 30 minutes for the 4 hour duration between muscle biopsies
  Other Names: Exercise Snacks
  Arms: Step-Reduction

SUMMARY:
The purpose of this study is to assess the impact of 3-days reduced physical activity (<1500 steps/day) with/without 'exercise snacks' (15 chair stands with calf raises every 30 min) on skeletal muscle metabolic health.

DETAILED DESCRIPTION:
Many adults gradually lose muscle size, strength, and function after the age of 50. These losses are believed to occur faster with periods of reduced activity (e.g., lower step counts or physical movement when sick or injured) and can be difficult to regain by merely returning to a previously normal activity status. Such periods of reduced activity can also impair the body's ability to use the nutrients in the food consumed (e.g., proteins and carbohydrates), which increases the risk of frailty, type 2 diabetes, and ultimately a reduced quality of life. It is important to identify strategies to prevent these losses in muscle size, strength, and function especially during periods of reduced activity.

Recently, our laboratory has found that performing repeated bodyweight chair squats (repeated sit-to-stands with a calf raise) during a single day of reduced activity improves the muscle's ability to use carbohydrates and proteins, which may be a viable strategy to offset the negative effects of step reduction on muscle health.

In this study, the investigators will assess whether completing bodyweight chair squats at regular intervals (i.e., 'exercise snacks') reduces the negative effects of step reduction on carbohydrate and protein metabolism following a meal. The investigators will determine the impact of 'exercise snacks' (15 chair stands with calf raises every 30 min) compared to seated rest on protein and carbohydrate metabolism following three days of step reduction. The investigators will also assess how these responses compare to those seen following three days of normal (i.e., habitual) activity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy older (age: 60-80 y) adults
* BMI between normal to overweight (18.5-29.9 kg/m2)

Exclusion Criteria:

* Regular use of nonsteroidal anti-inflammatory drugs (with the exception of daily low-dose aspirin)
* Alcohol consumption during the study period
* Use of anticoagulants
* Use of a walker, cane, or assistive walking device
* Current or recently remised cancer
* Infectious or gastrointestinal disease
* Inability to comply with study protocol (e.g., >1,500 steps/day during Step-Reduction Phase)
* Regular tobacco use
* Self-reported illicit drug use (e.g. growth hormone, testosterone, etc.)
* Diagnosed chronic illness (e.g. type 2 diabetes, heart disease, thyroid disease)
* Hormonal Replacement Therapy

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Myofibrillar protein synthesis rates | 5 Hours
  Myofibrillar protein synthesis rates assessed by incorporation of oral stable isotope tracer in both arms.

SECONDARY OUTCOMES:
Whole-body protein turnover | 5 Hours
  Whole-body protein turnover assessed by oral stable isotope tracers in both arms.
Amino acid oxidation and net protein balance | 5 Hours
  Amino acid oxidation and net protein balance assessed by oral tracers in both arms. Net protein balance is derived from the difference between amino acid intake (known) and total amino acid oxidation over the 5h measurement period.
Postprandial insulin area under the curve (AUC) to mixed macronutrient breakfast | 5 Hours postprandial
  The plasma insulin concentration measured by enzyme-linked immunosorbent assay (ELISA) area under the curve (AUC) will be quantified using the trapezoidal rule.
Postprandial glucose area under the curve (AUC) to mixed macronutrient breakfast | 5 hours postprandial
  The plasma glucose concentration measured by hexokinase method area under the curve (AUC) will be quantified using the trapezoidal rule.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel R Moore, PhD, Principal Investigator — University of Toronto; Hugo JW Fung, PhD, Study Director — University of Toronto
Locations (1):
- Goldring Center for High Performance Sport, Toronto, Ontario, Canada